CLINICAL TRIAL: NCT02071511
Title: Renal Denervation In Patient Undergoing VT Ablation:Combined Renal Denervation and VT Ablation vs. Simply VT Ablation
Acronym: ARDEVAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Sponsor appreciate the devastating impact that the results of the SYMPLICITY HTN 3 trial had on research progress for renal denervation. Based on the lack of recent progress, it is no longer practical to maintain the agreement.
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PV4286
Record Dates: First submitted 2014-02-10; First posted 2014-02-26 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Ventricular Tachycardia; Cardiomyopathy
MeSH Terms: conditions — Tachycardia, Ventricular; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Active Comparator): Ablation of ventricular arrhythmias
  Interventions: Procedure: Ablation of ventricular arrhythmias
- intervention group (Sham Comparator): Ablation of ventricular arrhythmias + renal denervation
  Interventions: Procedure: Ablation of ventricular arrhythmias + renal denervation

INTERVENTIONS:
Procedure: Ablation of ventricular arrhythmias — control group: Ablation of ventricular arrhythmias
  Arms: control group
Procedure: Ablation of ventricular arrhythmias + renal denervation — Intervention group: Ablation of ventricular arrhythmias + renal denervation
  Arms: intervention group

SUMMARY:
Study hypothesis:

With optimal medical therapy and repeated ablations, an additional renal denervation may have protective effects in terms of vegetative intrinsic activity and lead to a significant reduction in VT Burdens.

Study design:

Multicenter, randomized, prospective, single-blind clinical trial.

DETAILED DESCRIPTION:
Study protocol:

Catheter ablation of ventricular tachycardia versus combined catheter ablation of ventricular tachycardia and renal denervation.

A total of 50 patients with ventricular tachycardia treated with ICD shocks or ATP will be enrolled in this study. The randomization in the study is done before ablation.

For the ablation, an arterial access is required in both groups. During a 30 minutes waiting time which will apply to both groups, renal denervation will be performed.

In this period of time operators and staff will be blinded for the procedure, thereby they won't know if the patients will receive a renal denervation, in that way the investigators are avoiding a bias of future treatment of the patients.

Follow up and repeat procedures:

All Patients will be followed for a period of 3, 6, 9, 12 and 18 months after the procedure.

Regular visits are done in the investigators office. The visit will include ICD Interrogation, VT documentation in ICD Holter, 24-hour Holter ECG or Tele-ECGs, echocardiography.

Re- VT ablations are allowed at any time. In case of renal artery stenosis, denervation will not be performed. Drug therapy can be continued.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ischemic cardiomyopathy
* NYHA II-III
* Recurrent ventricular tachycardia, ICD interventions (shock or ATP)
* Obtained written informed consent

Exclusion Criteria:

* Age <18 years
* Previous VT ablation
* NYHA IV
* Cardiopulmonary decompensation within the last 4 weeks
* Pregnant women or women of childbearing potential without a negative pregnancy test within 48 hours prior to treatment
* History of hemorrhagic diathesis or other coagulopathies
* Contraindication for oral anticoagulation
* Hyper- or hypothyroidism
* Drug or chronic alcohol abuse
* Has any condition that would make participation not be in the best interest of the subject
* Incompliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Patients with adverse events such as recurrens of Ventricular Tachycardias or necessary Intracardiac shocks during 24 months follow up | 24 months
  Number of Patients with adverse events such as recurrens of Ventricular

SECONDARY OUTCOMES:
Number of Patients with Ventricular extrasystoles and non-sustained Ventricular Tachycardias compared to the time prior to ablation during 24 months follow up | 24 months
  Number of Patients with Ventricular extrasystoles and non-sustained Ventricular Tachycardias compared to the time prior to ablation during 24 months follow up
Number of periprocedural complications | 24 months
  Number of periprocedural complications

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Willems, MD, Principal Investigator — ASKLEPIOS St. Georg
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
We at Medtronic certainly appreciate the devastating impact that the results of the SYMPLICITY HTN 3 trial had on research progress for renal denervation, including your trial. Therefore, based on the lack of recent progress, it is no longer practical to maintain our agreement and we are hereby terminating our support for the trial.